CLINICAL TRIAL: NCT00573651
Title: Pilot Study of the Safety and Efficacy of Quadrivalent Human Papillomavirus Vaccine (Gardasil®) in Female Subjects With Juvenile Idiopathic Arthritis (JIA)/ Seronegative Arthritis
Brief Title: Safety and Efficacy of Gardasil in Females With Juvenile Idiopathic Arthritis (JIA)/Seronegative Arthritis
Acronym: CHASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); MetroHealth System, Ohio (Other); The Cleveland Clinic (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Nora G. Singer, M.D., MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Gardasil in JIA; CHASE (Other: UHClevelandMC)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-01

CONDITIONS: Arthritis
Keywords: JIA; SEA syndrome; AS; psoriatic arthritis; HPV vaccine
MeSH Terms: conditions — Arthritis; Arthritis, Psoriatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Open label vaccination study Gardasil vaccine (4 component).
Masking Description: The geometric mean titers are analyzed in a de-identified manner at Merck Contract laboratories.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JIA except SJIA with active systemic symptoms (Other): Females age 9-26 with JIA of all types that have had arthritis and do not have active systemic symptoms. All study subjects are receiving the Gardasil vaccine as part of their clinical care. The study observes outcomes related to this clinical care. Study intervention consists of some Blood Draws for serum titers taken to measure antibody.
  Interventions: Other: Blood Draws for Serum Titers

INTERVENTIONS:
Other: Blood Draws for Serum Titers — All study subjects are receiving the Gardasil vaccine as part of their clinical care. The Gardasil vaccine is not given because of study participation. The study observes outcomes related to this clinical care. Study intervention consists of some blood samples taken to measure antibody and RNA titers. Other study specific procedures performed include Questionnaires and observational data.

SUMMARY:
The purpose of this research study is to see if patients with juvenile idiopathic arthritis or seronegative arthritis (and related conditions) mount protective immune responses to the human papillomavirus (HPV) vaccine called Gardasil. The researchers also want to monitor for any increase in disease activity following receipt of the vaccine.

DETAILED DESCRIPTION:
Each individual subject's participation is scheduled to last approximately two years. Patients will be given Gardasil injections at months 0, 2, and 6. Patients will have geometric mean titers (GMT) measured at 7, 12, and 24 months. Questionnaires about health and function will also be completed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age 9-26 years, with polyarticular JIA, pauciarticular JIA, and sero-negative arthritis.

Exclusion Criteria:

* Pregnancy
* Known allergy/sensitivity or any hypersensitivity to yeast or components of study drug or their formulation
* Systemic onset JIA with active systemic symptoms (systemic onset JIA with polyarticular features but no fever or rash may be included).
* Prior vaccination against HPV
* Known HPV infection
* Current or history of cervical cancer or cervical intraepithelial neoplasia (CIN).

Males are excluded from this study because Gardasil® is currently approved only for females.

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2007-11; Primary Completion 2014-10-20 (Actual); Study Completion 2014-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nora G Singer, MD, Study Director — UHospitals Cleveland
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - University Hospitals Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from pediatric rheumatology clinics at UHCleveland Medical Center, Cleveland Clinic, the MetroHealth System, and the University of Chicago.
  Recruitment began in October of 2007 (IRB approval 10/22/2007) and finished in October of 2014.
Pre-assignment Details: This is open label vaccine on top of current therapy.
Groups:
- JIA Except SJIA Active Systemic Symptoms: Females age 9-26 with JIA of all types that have had arthritis and do not have active systemic symptoms. All study subjects are receiving the Gardasil vaccine as part of their clinical care. The study observes outcomes related to the clinical care. Study intervention consists of some Blood Draws for serum titers taken to measure antibody.
Period: Overall Study
Arm/Group | JIA Except SJIA Active Systemic Symptoms
Started (one patient withdrew consent) | 43
Completed (Any one who got a blood draw after the 3rd vaccine are considered completed as the primary outcome is available.) | 39
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Aggregate of All Three Arms.: All girls enrolled in the study 9-26 data were analyzed together as the original 72 subjects planned was not large enough to have statistically significant results once it became apparent that outcomes would need to be not only analyzed by subgroup but also by age 9-15 and 16-26.
Arm/Group | Aggregate of All Three Arms.
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Positive Serum GMTs at 7 Months (HPV06)
Description: dichotomized as negative or positive
Time Frame: 7 months
Population: 3 samples were lost in transport to lab
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 35
participants | 34

2. Primary Outcome: Positive Serum GMTs at 7 Months (HPV11)
Description: dichotomized as negative or positive
Time Frame: 7 months
Population: 3 samples were lost in transport to lab
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 35
participants | 35

3. Primary Outcome: Positive Serum GMTs at 7 Months (HPV16)
Description: dichotomized as negative or positive
Time Frame: 7 months
Population: 3 samples were lost in transport to lab
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 35
participants | 35

4. Primary Outcome: Positive Serum GMTs at 7 Months (HPV18)
Description: dichotomized as negative or positive
Time Frame: 7 months
Population: 3 samples were lost in transport to lab
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 35
participants | 35

5. Secondary Outcome: Disease Flare
Description: increased arthritis requiring addition of steroids, intensification of NSAIDs or new DMARD or biological DMARD
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 42
participants | 27

6. Secondary Outcome: Peds QL
Description: worsening of >30% from the prior visit
Time Frame: 2 years
Reporting Status: Not Posted

7. Secondary Outcome: Positive Serum GMT (HVP06)
Description: dichotomized as negative or positive
Time Frame: 12 months
Population: Not all participants agreed to blood draw, 2 missed visits and 2 drop outs.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 27
participants | 27

8. Secondary Outcome: Positive Serum GMT (HVP11)
Description: dichotomized as negative or positive
Time Frame: 12 months
Population: Not all participants agreed to blood draw, 2 missed visits and 2 drop outs.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 27
participants | 26

9. Secondary Outcome: Positive Serum GMT (HVP16)
Description: dichotomized as negative or positive
Time Frame: 12 months
Population: Not all participants agreed to blood draw, 2 missed visits and 2 drop outs.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 27
participants | 27

10. Secondary Outcome: Positive Serum GMT (HVP18)
Description: dichotomized as negative or positive
Time Frame: 12 months
Population: Not all participants agreed to blood draw, 2 missed visits and 2 drop outs.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 27
participants | 27

11. Secondary Outcome: Positive Serum GMT (HPV06)
Time Frame: 24 months
Population: Not all participants agreed blood draw, and subject withdraw.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 12
participants | 11

12. Secondary Outcome: Positive Serum GMT (HPV11)
Time Frame: 24 months
Population: Not all participants agreed blood draw, and subject withdraw.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 12
participants | 9

13. Secondary Outcome: Positive Serum GMT (HPV16)
Time Frame: 24 months
Population: Not all participants agreed blood draw, and subject withdraw.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 12
participants | 11

14. Secondary Outcome: Positive Serum GMT (HPV18)
Time Frame: 24 months
Population: Not all participants agreed blood draw, and subject withdraw.
Measure: Number; unit: participants
Arm/Group | JIA Except SJIA With Active Systemic Symptoms
Number analyzed (Participants) | 12
participants | 8

ADVERSE EVENTS:
Time Frame: Data was collected for up to completion of the 24 month visit for patients that completed the study or the last known study visit.
Description: In the initial protocol pregnancy after immunization was not excluded as an SAE. The label for Gardasil vaccine however does not say that patients need to avoid pregnancy following the immunization series. We had one pregnancy during the follow up period. The IRB protocol was amended to exclude pregnancy as an SAE once all vaccines are complete during the follow up period.
Arm/Group | Aggregate of All Three Arms.
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 1/43
Other Adverse Events (participants affected / at risk) | 21/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggregate of All Three Arms. (N=43)
pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) — This pregnancy occurred months after the immunization series was completed.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggregate of All Three Arms. (N=43)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 10 (11) — Sinusitis, cold, cough
Achiness (Infections and infestations) | 3 (3) — fatigue/flu-like symptoms
nausea or diarrhea (Gastrointestinal disorders) | 8 (8) — stomach upset
arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) — stiffness
lightheadedness (Vascular disorders) | 5 (5) — dizziness
fever (Infections and infestations) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 1 (2) — urticaria
bruise (Musculoskeletal and connective tissue disorders) | 2 (3) — contusion
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
strep throat (Infections and infestations) | 2 (2)
syncope vaso-vagal (Vascular disorders) | 1 (1)
flare (Musculoskeletal and connective tissue disorders) | 2 (2) — arthritis flare, enthesitis flare
dry socket following extraction (Injury, poisoning and procedural complications) | 1 (1) — complications wisdom tooth extraction
otalgia (Ear and labyrinth disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) — Shingles
Injection site pain (Injury, poisoning and procedural complications) | 1 (1) — injection șite reaction
insomnia (General disorders) | 1 (1) — sleep disorder
musculoskeletal pain due to MVA injury (Injury, poisoning and procedural complications) | 1 (1) — joint pain due to car accident
warts, plantar (Infections and infestations) | 1 (1)
thrush (Infections and infestations) | 1 (1) — oral candidiasis
vomiting (Gastrointestinal disorders) | 2 (2) — emesis, stomach flu

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No